CLINICAL TRIAL: NCT04949100
Title: Microcurrent for Fibromyalgia, a Double-Blinded, Placebo-Controlled Study
Brief Title: Microcurrent for Fibromyalgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Crawford (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20210098H
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: chronic pain; microcurrent
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Microcurrent (Experimental)
  Interventions: Device: Microcurrent Transcutaneous Electrical Nerve Stimulator (TENS) for pain relief
- Placebo (Placebo Comparator)
  Interventions: Device: PLACEBO Microcurrent Transcutaneous Electrical Nerve Stimulator (TENS) for pain relief

INTERVENTIONS:
Device: Microcurrent Transcutaneous Electrical Nerve Stimulator (TENS) for pain relief — * Duration: 60 minutes.
  * Electrode placement: There will be one lead placed on the back of the neck and one placed on lower abdomen.
  * Frequency: Each lead delivers a dual channel microcurrent of 10 and 40 Hz simultaneously.
  * Amperage: Adjusted according to BMI: 100 μA for an underweight BMI less 20, 300μA for an overweight BMI greater than 30, and 200μA for normal BMI (20-30). Amperage may be adjusted to 20-300 μA according to comfort.
  * Positioning: The patient remains seated for the first 10 minutes with the investigator watching for any side effects. The patient may stand, sit, lie supine, et cetera for the remainder of treatment.
  Arms: Microcurrent
Device: PLACEBO Microcurrent Transcutaneous Electrical Nerve Stimulator (TENS) for pain relief — * Duration: 60 minutes.
  * Frequency: None
  * Electrode placement: There will be one lead placed on the back of the neck and one placed on lower abdomen.
  * Amperage: None
  * Positioning: The patient remains seated for the first 10 minutes, again, with the investigator watching for any side effects. The patient may stand, sit, lie supine, et cetera for the remainder of treatment.
  Arms: Placebo

SUMMARY:
Explore the use of microcurrent therapy for fibromyalgia patients and evaluate its effect on generalized pain and quality of life.

Determine if microcurrent therapy be effectively self-administered by the patient as an adjunct to medical pain management.

DETAILED DESCRIPTION:
This study is not intended to be definitive and should be considered an exploratory randomized trial to determine conditions for which microcurrent is more effective. Thus, extensive subgroup analyses will be performed so that definitive trials can be developed. This is a double-blind study where subjects will not know if they are receiving microcurrent treatment.

Day 0, Screening visit (may occur during the patient's regular health visit):

* Obtain and document signed Informed Consent document and HIPAA Authorization.
* Review past medical history to verify inclusion/exclusion criteria.
* Proper hydration is essential before any microcurrent therapy. Hydration is ensured by the patient drinking at least 8 ounces of water 1 hour before treatment.
* Record onset and chronicity of fibromyalgia syndrome
* Record any medicines that the subject is taking.
* Collect demographic information to include age, weight (pounds), height (inches), race, ethnicity, and sex.
* Record any standard treatment subject is receiving. Standard treatment may include, but is not limited to one or more of the following: medications, physical therapy, acupuncture, pain management clinic, dry needling, occupational therapy, osteopathic manipulative treatment,

Randomization: Subjects will be randomized using complete block design with repeated measure into one of two research-related treatment groups: Group 1 (microcurrent) and Group 2 (placebo microcurrent)

Day 1 (may be same day as screening):

* Subjects will complete the following pre-treatment:

  * Measure Yourself Medical Outcome Profile (MYMOP)
  * Revised Fibromyalgia Impact Questionnaire (FIQR)
* Pre-treatment measurement of active range of motion of both wrists, knees, trunk, neck, and head with the Myovision 3G Wireless System (Myovision, Seattle, WA) ¹ .

  --*(Myovision will be performed for some subjects based off the availability of Myvision trained staff)
* Proper hydration is essential before any microcurrent therapy. Hydration is ensured by the patient drinking at least 8 ounces of water 1 hour before treatment.
* Research participant will receive microcurrent according to their randomization group.
* Post-treatment measurement of active range of motion of both wrists, knees, trunk, neck, and head with the Myovision 3G Wireless System (Myovision, Seattle, WA) ¹ .
* Research participant will be loaned a microcurrent box to bring home with them for this study. They will be instructed to bring the microcurrent box back. A hand-receipt will be signed by the patient accepting responsibility for device replacement if they fail to return or break it.

Day 2-7 (at home microcurrent application):

-The research participant will self-administer the microcurrent according to their randomization group daily.

Day 8:

* Subjects will complete the following pre-treatment:

  * MYMOP
  * Revised Fibromyalgia Impact Questionnaire (FIQR)
* Pre-treatment measurement of active range of motion of both wrists, knees, trunk, neck, and head with the Myovision 3G Wireless System (Myovision, Seattle, WA) ¹ .

  --*(Myovision will be performed for some subjects based off the availability of Myvision trained staff)
* Proper hydration is essential before any microcurrent therapy. Hydration is ensured by the patient drinking at least 8 ounces of water 1 hour before treatment.
* Research participant will receive microcurrent according to their randomization group.
* Post-treatment measurement of active range of motion of both wrists, knees, trunk, neck, and head with the Myovision 3G Wireless System (Myovision, Seattle, WA) ¹ .

Day 15 Final Visit:

* Subjects will complete the following:

  * MYMOP
  * Revised Fibromyalgia Impact Questionnaire (FIQR)
* Measurement of active range of motion of both wrists, knees, trunk, neck, and head with the Myovision 3G Wireless System (Myovision, Seattle, WA) ¹ . --*(Myovision will be performed for some subjects based off the availability of Myvision trained staff)

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female Active Duty or DoD beneficiary aged 18-74 years old.
* Meets diagnostic criteria of fibromyalgia as defined by the American College of Rheumatology 1990 Criteria 1,18 to be consistent with prior research.
* Symptom duration of at least 3 months
* Tender points: having >10/18 tender points
* Pain-affected areas includes all quadrants of the body
* Other causes excluded clinically
* History of a neck injury sometime in their life

Exclusion Criteria:

* Peripheral neuropathy
* Pregnancy
* History of:

  * Brain/spine surgery
  * Nerve entrapment surgery
  * Severe bony deformities or contracture
  * Hypersensitive reaction to the surface electrode
  * Severe psychological disorders
  * Current alcohol or drug abuse. (caveat: medical marijuana is permitted)
* Active infections
* Active cancer
* Cardiac arrhythmias (If yes, please list _____________)
* Received an organ transplant
* Pacemakers and electrically implanted electronic devices
* Subjects scheduled for surgery will not be eligible to participate in thisstudy until 6 weeks post-surgery.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Day 1
  The FIQR assesses three domains (function, overall impact and symptoms) from which a total score of pain impact is derived. FMS patients have a mean (SD) total score of 56.6 (19.9) and healthy patients have a mean (SD) total score of 12.1 (11.6). FMS patients' means for function, overall impact and symptoms domains are 15.6, 11.0, and 30.0 respectively. Higher total scores are indicative of greater dysfunction or symptom severity. While total scores are slightly negatively skewed favoring severe cases, scores can be assessed with parametric methods.
Revised Fibromyalgia Impact Questionnaire (FIQR) | Day 8
  The FIQR assesses three domains (function, overall impact and symptoms) from which a total score of pain impact is derived. FMS patients have a mean (SD) total score of 56.6 (19.9) and healthy patients have a mean (SD) total score of 12.1 (11.6). FMS patients' means for function, overall impact and symptoms domains are 15.6, 11.0, and 30.0 respectively. Higher total scores are indicative of greater dysfunction or symptom severity. While total scores are slightly negatively skewed favoring severe cases, scores can be assessed with parametric methods.
Revised Fibromyalgia Impact Questionnaire (FIQR) | Day 15
  The FIQR assesses three domains (function, overall impact and symptoms) from which a total score of pain impact is derived. FMS patients have a mean (SD) total score of 56.6 (19.9) and healthy patients have a mean (SD) total score of 12.1 (11.6). FMS patients' means for function, overall impact and symptoms domains are 15.6, 11.0, and 30.0 respectively. Higher total scores are indicative of greater dysfunction or symptom severity. While total scores are slightly negatively skewed favoring severe cases, scores can be assessed with parametric methods.
Measure Yourself Medical Outcome Profile (MYMOP) | Day 1
  The MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1. The MYMOP scales are ordinal and will be assess with nonparametric methods.
Measure Yourself Medical Outcome Profile (MYMOP) | Day 8
  The MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1. The MYMOP scales are ordinal and will be assess with nonparametric methods.
Measure Yourself Medical Outcome Profile (MYMOP) | Day 15
  The MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1. The MYMOP scales are ordinal and will be assess with nonparametric methods.
active range of motion (AROM) | day 1 immediately pre-treatment
  AROM (degrees) will be measured for both wrists, knees, trunk, neck, and head using the Myovision 3G Wireless System. The data is interval and will be assessed with parametric methods.
  MyoVision System: MyoVision DynaROM (Dynamic Range Of Motion) is a functional and objective soft tissue injury test that measures muscle guarding and range of motion by assessing both while a patient moves. Data is sent to computer software and graphed for interpretation. DynaROM is FDA cleared, class II diagnostic equipment.
  *(Myovision will be performed for some subjects based off the availability of Myvision trained staff)*
active range of motion (AROM) | day 1 immediately post-treatment
  AROM (degrees) will be measured for both wrists, knees, trunk, neck, and head using the Myovision 3G Wireless System. The data is interval and will be assessed with parametric methods.
  MyoVision System: MyoVision DynaROM (Dynamic Range Of Motion) is a functional and objective soft tissue injury test that measures muscle guarding and range of motion by assessing both while a patient moves. Data is sent to computer software and graphed for interpretation. DynaROM is FDA cleared, class II diagnostic equipment.
  *(Myovision will be performed for some subjects based off the availability of Myvision trained staff)*
active range of motion (AROM) | day 8
  AROM (degrees) will be measured for both wrists, knees, trunk, neck, and head using the Myovision 3G Wireless System. The data is interval and will be assessed with parametric methods.
  MyoVision System: MyoVision DynaROM (Dynamic Range Of Motion) is a functional and objective soft tissue injury test that measures muscle guarding and range of motion by assessing both while a patient moves. Data is sent to computer software and graphed for interpretation. DynaROM is FDA cleared, class II diagnostic equipment.
  *(Myovision will be performed for some subjects based off the availability of Myvision trained staff)*
active range of motion (AROM) | day 15
  AROM (degrees) will be measured for both wrists, knees, trunk, neck, and head using the Myovision 3G Wireless System. The data is interval and will be assessed with parametric methods.
  MyoVision System: MyoVision DynaROM (Dynamic Range Of Motion) is a functional and objective soft tissue injury test that measures muscle guarding and range of motion by assessing both while a patient moves. Data is sent to computer software and graphed for interpretation. DynaROM is FDA cleared, class II diagnostic equipment.
  *(Myovision will be performed for some subjects based off the availability of Myvision trained staff)*

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Sprott H. What can rehabilitation interventions achieve in patients with primary fibromyalgia? Curr Opin Rheumatol. 2003 Mar;15(2):145-50. doi: 10.1097/00002281-200303000-00011. PMID 12598803
- [Background] Lempp HK, Hatch SL, Carville SF, Choy EH. Patients' experiences of living with and receiving treatment for fibromyalgia syndrome: a qualitative study. BMC Musculoskelet Disord. 2009 Oct 7;10:124. doi: 10.1186/1471-2474-10-124. PMID 19811630
- [Background] Rossy LA, Buckelew SP, Dorr N, Hagglund KJ, Thayer JF, McIntosh MJ, Hewett JE, Johnson JC. A meta-analysis of fibromyalgia treatment interventions. Ann Behav Med. 1999 Spring;21(2):180-91. doi: 10.1007/BF02908299. PMID 10499139
- [Background] Bertolucci LE, Grey T. Clinical comparative study of microcurrent electrical stimulation to mid-laser and placebo treatment in degenerative joint disease of the temporomandibular joint. Cranio. 1995 Apr;13(2):116-20. doi: 10.1080/08869634.1995.11678054. PMID 8697497
- [Background] McMakin: Frequency Specific Microcurrent in Pain Management, Textbook for practitioners. Edinburgh: Elsevier Science Press, 2010
- [Background] Cheng N, Van Hoof H, Bockx E, Hoogmartens MJ, Mulier JC, De Dijcker FJ, Sansen WM, De Loecker W. The effects of electric currents on ATP generation, protein synthesis, and membrane transport of rat skin. Clin Orthop Relat Res. 1982 Nov-Dec;(171):264-72. PMID 7140077
- [Background] Salvat I, Zaldivar P, Monterde S, Montull S, Miralles I, Castel A. Functional status, physical activity level, and exercise regularity in patients with fibromyalgia after Multidisciplinary treatment: retrospective analysis of a randomized controlled trial. Rheumatol Int. 2017 Mar;37(3):377-387. doi: 10.1007/s00296-016-3597-x. Epub 2016 Nov 14. PMID 27844124
- [Background] McMakin CR, Oschman JL. Visceral and somatic disorders: tissue softening with frequency-specific microcurrent. J Altern Complement Med. 2013 Feb;19(2):170-7. doi: 10.1089/acm.2012.0384. Epub 2012 Jul 9. PMID 22775307
- [Background] Curtis D, Fallows S, Morris M, McMakin C. The efficacy of frequency specific microcurrent therapy on delayed onset muscle soreness. J Bodyw Mov Ther. 2010 Jul;14(3):272-9. doi: 10.1016/j.jbmt.2010.01.009. Epub 2010 Feb 19. PMID 20538225
- [Background] McMakin, C.: Cytokine changes with microcurrent treatment of fibromyalgia. Journal of Bodywork and Movement Therapies, 9: 169, 2005
- [Background] Hewlett, K.: Microcurrent treatment on pain, edema, and decreased muscle force associated with delayed onset muscle soreness: a double-blind, placebo, study. In: Kinesiology & Leisure Sciences: University of Hawaii at Manoa, 2003
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Background] Day A. The development of the MYMOP pictorial version. Acupunct Med. 2004 Jun;22(2):68-71. doi: 10.1136/aim.22.2.68. PMID 15253581
- [Background] Paterson C, Britten N. In pursuit of patient-centred outcomes: a qualitative evaluation of the 'Measure Yourself Medical Outcome Profile'. J Health Serv Res Policy. 2000 Jan;5(1):27-36. doi: 10.1177/135581960000500108. PMID 10787584
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Hauser W, Wolfe F. Diagnosis and diagnostic tests for fibromyalgia (syndrome). Reumatismo. 2012 Sep 28;64(4):194-205. doi: 10.4081/reumatismo.2012.194. PMID 23024964
- [Background] Gerhardt J., Cocchiarella L., Lea R. The practical guide to range of motion assessment. American Medical Association; Chicago: 2001. pp. 25-32.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Lehman, Eric L. (2006). Nonparametrics: Statistical Methods Based on Ranks, Revised, pages 76-81.
- [Background] Holm, S. 1979. A simple sequential rejective multiple test procedure. Scand. J. Statistics, 6: 65-70
- [Background] R Core Team (2014). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL http://www.R-project.org/.